CLINICAL TRIAL: NCT01057238
Title: Intensive Communication for Chronically Critically Ill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Barbara J. Daly, Principal Investigator, Case Western Reserve University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01NR008941 (NIH)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Critical Care
Keywords: mechanical ventilation; critical care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Communication (Experimental): regular family meeting every 5 days.
  Interventions: Other: Intensive Communication System
- Control (No Intervention): usual care

INTERVENTIONS:
Other: Intensive Communication System — Regular family meetings once a week, using a standard protocol
  Other Names: Intervention arm
  Arms: Intensive Communication

SUMMARY:
This study was a trial of a formal system of family meetings to support family decision makers of chronically critically ill patients in the intensive care unit.

DETAILED DESCRIPTION:
Formal family meetings have been recommended as a useful approach to assist in goal setting, facilitate decision making, and reduce use of ineffective resources in the ICU. We implemented an "intensive communication system" to test the effect of regular, structured formal family meetings on patient outcomes among long-stay ICU patients

The design was a pre-post, tandem assignment of patients (n=217) receiving usual care and communication, followed by enrollment of intervention patients (n=354), from 5 ICUs. The "intensive communication system" included: (1) family meeting within 5 days of ICU admission and weekly thereafter; (2) each meeting addressed medical update, values and preferences, goals of care; treatment plan, and milestones for judging effectiveness of treatment.

We measured differences between control and intervention patients in indicators of aggressiveness of care or timing of treatment limitation decisions (ICU mortality, LOS, duration of ventilation, treatment limitation orders, or use of tracheostomy or percutaneous gastrostomy). Difference in outcomes among patients who died or who had treatment limitation orders, comparing control and intervention groups, was also examined.

ELIGIBILITY:
Inclusion Criteria:

* cognitively impaired mechanical ventilation >3 days not expected to be discharged before 5 days having a family decision maker

Exclusion Criteria:

* no family member hospice referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
length of stay and depression | ICU admission, Day 5, discharge, and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Daly, PhD, RN, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hosptials Case Medical center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Daly BJ, Douglas SL, O'Toole E, Gordon NH, Hejal R, Peerless J, Rowbottom J, Garland A, Lilly C, Wiencek C, Hickman R. Effectiveness trial of an intensive communication structure for families of long-stay ICU patients. Chest. 2010 Dec;138(6):1340-8. doi: 10.1378/chest.10-0292. Epub 2010 Jun 24. PMID 20576734